CLINICAL TRIAL: NCT00977470
Title: Phase II Study of Erlotinib With or Without Hydroxychloroquine in Patients With Previously Untreated Advanced NSCLC and EGFR Mutations
Brief Title: Erlotinib With or Without Hydroxychloroquine in Chemo-Naive Advanced NSCLC and (EGFR) Mutations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stanford University (Other); Yale University (Other); University of Maryland (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Lecia V. Sequist, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-097; OSI4620s (Other: OSI)
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; HCQ; erlotinib; Tarceva
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib (Experimental): Erlotinib 150 mg oral daily
  Interventions: Drug: Erlotinib
- Erlotinib and Hydroxychloroquine (Experimental): Erlotinib 150 mg oral daily plus Hydroxychloroquine (HCQ) 1000 mg oral daily
  Interventions: Drug: Erlotinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Erlotinib — 150 mg taken orally once daily
  Other Names: Tarceva
Drug: Hydroxychloroquine — 1000 mg taken orally once daily after erlotinib
  Other Names: HCQ
  Arms: Erlotinib and Hydroxychloroquine

SUMMARY:
The purpose of this research study is to learn if adding hydroxychloroquine (HCQ) to erlotinib helps treat non-small cell lung cancer (NSCLC). Another goal of this research study is to learn more about NSCLC and how it may respond to study treatment. Erlotinib (Tarceva) is a type of drug called a tyrosine kinase inhibitor (TKI). TKIs block a protein called the epidermal growth factor receptor (EGFR). EGFR may control tumor growth and tumor cell survival. However, although TKI drugs can work for some lung cancer patients for a period of time, eventually the tumor finds a way to resist or counteract the TKI treatment and it begins to grow again. Hydroxychloroquine (HCQ) is a drug approved by the FDA for treating malaria, rheumatoid arthritis, and several other diseases. Laboratory research suggests that when HCQ is given with a TKI, it may help delay or prevent TKI resistance from developing.

DETAILED DESCRIPTION:
* Because no one knows which of the study options are best, participants will be randomized into of the study groups: Group A (erlotinib) or Group B (erlotinib and HCQ). Study treatment will be divided into time periods called cycles. Each study treatment cycle is 28 days.
* Erlotinib (Group A and Group B) will be taken orally once a day. Hydroxychloroquine (Group B) will be taken orally once a day after taking erlotinib.
* The following tests and procedures will be performed day 1 of each cycle: physical examination, performance status assessment, questions about any symptoms or side effects, blood for routine tests. The following procedures will be performed at certain study visits: Research blood tests (cycle 1, cycle 2, then every other even cycle); eye exam (cycle 4, cycle 7, and then every 3 months); assessment of the tumor with CT or MRI scan (done at the end of even cycles.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of non-small cell lung cancer
* Stage IV disease by the American Joint Committee on Cancer/IASLC 7th edition proposed edition staging criteria
* An EGFR sensitizing mutation must be detected in tumor tissue. Specifically, patients harboring the most common mutations, deletions in exon 19 or the L858R mutation in exon 21 are eligible. Presence of the known resistance mutation T790M as detected by direct tumor sequencing is not allowed. Other rare EGFR mutations may be eligible after discussion with the overall principal investigator
* Age equal to or greater than 18 years
* Measurable disease by RECIST criteria, defined as the presence of at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 10mm or greater with spiral CT scan
* ECOG Performance status of 0, 1 or 2
* Since prior radiation or surgery, 14 days or more must have elapsed before starting protocol treatment
* No prior treatment with erlotinib, gefitinib, or other small molecule EGFR-TKIs. Prior treatment in the adjuvant setting is allowed if at least 1 year has elapsed since TKI course.
* Adequate organ function as outlined in the protocol
* Patients must undergo a screening eye exam to obtain approval for HCQ treatment, which establishes the absence of baseline conditions include macular degeneration, visual field changes, other retinal disease, and cataracts that interfere with required funduscopic examinations
* No G6PD deficiency, as HCQ may cause hemolysis in patients with G6DP

Exclusion Criteria:

* Symptomatic CNS metastases or newly diagnosed CNS metastases that have not yet been definitively treated with radiation and/or surgery. Note that patients with a history of CNS metastases or cord compression are allowed if they have been definitively treated and are clinically stable. Maintenance steroids are allowed but maintenance seizure medication with an EIAED is not allowed
* Prior radiation therapy inclusive of all identified target lesions. Note that prior palliative radiation to bony disease, CNS disease, or a limited thoracic area is allowed, provided that there is measurable disease outside the field and radiation is completed at least two weeks prior to starting treatment and the patient has fully recovered from all side effects
* Current use of hydroxychloroquine for any reason
* Known hypersensitivity to chloroquine, hydroxychloroquine, or any closely related drug: erlotinib, gefitinib, or any closely related drug
* Patients who are pregnant or breastfeeding. Female subjects of childbearing potential and male subjects must practice acceptable methods of birth control
* Any evidence of clinically active interstitial lung disease. Note that patients with chronic, stable radiographic changes who are asymptomatic are eligible
* Invasive malignancies within the past 3 years except for adequately treated carcinoma of the cervix, basal or squamous cell carcinomas of the skin
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study, including a prior diagnosis of porphyria or non-light-sensitive psoriasis, as HCQ can significantly exacerbate both of these conditions
* Use of any non-FDA approved or investigational agent in 30 days or less of enrolling onto the trial, or failure to recover from the side effects of any of these agents
* Penicillamine use for Wilson's disease or any other indication, as concomitant use with HCQ can increase toxicity to penicillamine
* Life expectancy of less than 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-10; Primary Completion 2015-05 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia Sequist, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Stanford Cancer Institute, Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arvold ND, Heidari P, Kunawudhi A, Sequist LV, Mahmood U. Tumor Hypoxia Response After Targeted Therapy in EGFR-Mutant Non-Small Cell Lung Cancer: Proof of Concept for FMISO-PET. Technol Cancer Res Treat. 2016 Apr;15(2):234-42. doi: 10.1177/1533034615574386. Epub 2015 Mar 10. PMID 25759424

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Started | 38 | 38
Completed | 0 | 0
Not Completed | 38 | 38
Not completed — Lack of Efficacy | 32 | 30
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 0 | 2
Not completed — clinical decline | 0 | 1
Not completed — prolonged recovery post-surgery | 0 | 1
Not completed — Still on-study | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Median (Full Range); unit: years] | 63 [43 to 84] | 65 [37 to 82] | 64 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 14 | 15 | 29
Smoking History [Count of Participants; unit: Participants]
  Never smoked | 28 | 20 | 48
  <= 10 pack years | 4 | 8 | 12
  > 10 pack years/current | 6 | 10 | 16
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 33 | 31 | 64
  Non-small cell lung cancer, Not Otherwise Specifie | 5 | 7 | 12
Brain metastases [Count of Participants; unit: Participants] | 11 | 16 | 27
Prior chemotherapy [Count of Participants; unit: Participants] | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival
Description: A measure of progression-free survival in patients with advanced non small-cell lung cancer (NSCLC) and EGFR mutations treated with erlotinib as compared with patients treated with erlotinib plus hydroxychloroquine (HCQ). Disease progression is defined as at least a 20% increase in the sum of the longest diameter of target lesions, as seen on CT scan, or the appearance of one or more new lesions on CT scan.
Time Frame: From start of treatment until report of disease progression, assessed up to 10 years.
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Number analyzed (Participants) | 38 | 38
months | 10.8 [9.0 to 13.6] | 10.8 [7.0 to 14.6]

2. Primary Outcome: Nine-month Progression-free Survival Rate
Description: This trial can detect a difference in proportions alive without progression at 9 months from 50% in the erlotinib arm to 77% in the erlotinib plus hydroxychloroquine (HCQ) arm, using an alpha of 0.15 and power of 85%, using the two-sided Likelihood Ratio test. Progression is defined as at least a 20% increase in the size of existing lesions or the appearance of one or more new lesions.
Time Frame: Nine months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Number analyzed (Participants) | 38 | 38
percentage of participants | 71 [53 to 83] | 52 [35 to 67]
Statistical Analysis 1: Comparison: Erlotinib vs Erlotinib and Hydroxychloroquine; Test type: Equivalence — All enrolled patients will be included in the intent-to-treat efficacy analyses. Based on historical patients with EGFR mutations treated with gefitinib, we expect median progression-free survival on the erlotinib-alone arm to be approximately 9 months. This trial can detect a difference in proportions alive without progression at 9 months from 50% in the erlotinib arm to 77% in the erlotinib plus HCQ arm, using an alpha of 0.15 and power of 85%, using the two-sided Likelihood Ratio test; p = 0.28, Log Rank

3. Secondary Outcome: Treatment Related Toxicity, > 10% Frequency, Any Grade
Description: To evaluate the safety of treatment with erlotinib with and without hydroxychloroquine (HCQ). All participants receiving study treatment were evaluated for safety. Parameters included laboratory tests, hematological abnormalities, physical exam findings and spontaneous reports of adverse events reported by participants. Toxicities were evaluated and graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = fatal.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Number analyzed (Participants) | 38 | 38
Participants
  Diarrhea | 30 | 32
  Rash | 17 | 21
  Fatigue | 15 | 21
  Grade 3 Fatigue | 1 | 7
  Nausea | 11 | 21
  Anorexia | 9 | 11
  Taste changes | 9 | 9
  Grade 3 Taste changes | 0 | 1
  Alopecia | 5 | 7
  Weight loss | 5 | 7
  Ocular toxicity | 6 | 4
  Grade 4 or 5 events | 0 | 0

4. Secondary Outcome: Objective Tumor Response Rate Following Treatment With Erlotinib and With Erlotinib/HCQ.
Description: Response is assessed via spiral CT scan, done at baseline and after every 2 cycles of study treatment. Standard RECIST (Response Evaluation Criteria in Solid Tumors) was used. Complete Response (CR) = disappearance of all target lesions; Partial Response (PR) = at least a 30% decrease in the size of target lesions, as compared to baseline; Progressive Disease (PD) = at least at 20% increase in the size of target lesions, or the appearance of one or more new lesions; Stable Disease (SD) = neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
  Response rate = CR + PR. Disease control rate = CR + PR + SD
Time Frame: 2 years
Population: 1 participant in each arm (2 participants total) did not have any scans done after baseline and therefore response could not be assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Number analyzed (Participants) | 37 | 37
Participants
  Complete Response | 1 | 2
  Partial Response | 23 | 19
  Stable Disease | 10 | 10
  Progressive Disease | 3 | 6
  Response Rate | 24 | 21
  Disease Control Rate | 34 | 31

5. Secondary Outcome: Overall Survival of Patients Treated With Erlotinib and With Erlotinib/HCQ
Time Frame: Until death
Reporting Status: Not Posted, anticipated posting 2027-12

6. Other Pre Specified Outcome: Circulating Tumor Cell Quantification
Description: Serial circulating tumor cell (CTC) analyses will be performed on peripheral blood and correlated with disease response.
Time Frame: Until disease progression (median of 10.8 months)
Population: Due to technical reasons, this assay was not ready and therefore circulating tumor cell analysis was not done.
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: EGFR Mutational Status
Description: Correlation of molecular and genetic tumor characteristics with disease response. Genomic DNA will be extracted from tumor tissue and direct sequencing analysis will be performed to identify additional mutations.
Time Frame: 2 years
Population: Tumor tissue analysis was not performed for this correlative outcome.
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Percent of Participants in Which FMISO-PET ([18F]-Fluoromisonidazole-positron Emission Tomography) is Able to Detect and Quantify Changes in Tumor Hypoxia After Erlotinib.
Description: [18F]-FMISO-PET/CT was performed on a 64-slice PET/CT scanner and tracer uptake was assessed using SUV (standardized uptake value), normalizing the radioactivity measured in tissue by the injected dose and the body weight of the patient. Mean and maximum SUV and threshold volume of FMISO uptake were measured to quantify the extent of hypoxia in the primary tumor. Imaging was performed before and after initiation of therapy with erlotinib.
Time Frame: 12 weeks
Population: Only 2 participants were enrolled in this pilot companion study
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Number analyzed (Participants) | 2 | 0
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were collected via physical exam, eye exam and laboratory test. Additionally, participants were questioned at each study visit regarding other events not collected by the above methods.
Arm/Group | Erlotinib | Erlotinib and Hydroxychloroquine
Serious Adverse Events (participants affected / at risk) | 4/38 | 2/38
Other Adverse Events (participants affected / at risk) | 38/38 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=38) | Erlotinib and Hydroxychloroquine (N=38)
Pulmonary embolism (Vascular disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection, nos (Infections and infestations) | 0 | 1
Constitutional disorders - other (General disorders) | 1 | 0 — Failure to Thrive
Skin - pain (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Respiratory - other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Pneumomediastinum
Death NOS (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=38) | Erlotinib and Hydroxychloroquine (N=38)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Allergy-other (Immune system disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing-other (Ear and labyrinth disorders) | 1 (1) | 2 (3)
Hemoglobin (Investigations) | 4 (6) | 1 (3)
Leukocytes (Blood and lymphatic system disorders) | 1 (1) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4) | 2 (6)
Neutrophils (Blood and lymphatic system disorders) | 1 (3) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Hematologic-other (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia-other (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 10 (10) | 6 (6)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)
Cardiac-other (Cardiac disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 25 (32) | 27 (44)
Fever w/o neutropenia (General disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 10 (10)
Rigors/chills (General disorders) | 4 (4) | 2 (3)
Sweating (General disorders) | 0 (0) | 1 (1)
Weight loss (Investigations) | 7 (8) | 8 (9)
Constitutional, other (General disorders) | 5 (5) | 1 (1)
INR (Investigations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Chelitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (18) | 12 (13)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (7) | 10 (10)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 20 (31) | 13 (18)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 18 (25) | 21 (28)
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin-other (Skin and subcutaneous tissue disorders) | 20 (25) | 8 (10)
ADH secretion abnormality (eg SIADH) (Investigations) | 1 (1) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyopthyroidism (Endocrine disorders) | 3 (3) | 0 (0)
Endocrine-other (Endocrine disorders) | 1 (1) | 0 (0)
Growth and Development, Other (General disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 13 (15) | 15 (23)
Constipation (Gastrointestinal disorders) | 12 (13) | 11 (12)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 5 (6)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 33 (43) | 32 (44)
Distention/bloating, abdominal (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 5 (7)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (7) | 7 (7)
Hemorrhoids (Gastrointestinal disorders) | 3 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muco/stomatitis by exam, anus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 (2) | 1 (1)
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2 (2) | 1 (1)
Muco/stomatitis (symptom) pharynx (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (22) | 23 (38)
Taste disturbance (Gastrointestinal disorders) | 10 (11) | 10 (14)
Vomiting (Gastrointestinal disorders) | 7 (8) | 9 (10)
GI-other (Gastrointestinal disorders) | 1 (1) | 7 (9)
Anus, hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vagina, hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Lung, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hemorrhage-other (General disorders) | 2 (2) | 1 (1)
Infection w/ gr3-4 neut, ungual (nails) (Infections and infestations) | 1 (3) | 0 (0)
Infection Gr0-2 neut, bladder (Infections and infestations) | 1 (1) | 0 (0)
Infection Gr0-2 neut, bronchus (Infections and infestations) | 1 (1) | 0 (0)
Infection Gr0-2 neut, lung (Infections and infestations) | 1 (1) | 0 (0)
Infection Gr0-2 neut, skin (Infections and infestations) | 2 (2) | 0 (0)
Infection Gr0-2 neut, ungual (Infections and infestations) | 3 (5) | 3 (3)
Infection Gr0-2 neut, upper airway (Infections and infestations) | 4 (4) | 5 (5)
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 4 (5) | 4 (5)
Infection Gr0-2 neut, vagina (Infections and infestations) | 0 (0) | 1 (1)
Infection Gr0-2 neut, wound (Infections and infestations) | 0 (0) | 1 (1)
Infection w/ unk ANC eye NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection w/ unk ANC joint (Infections and infestations) | 2 (2) | 0 (0)
Infection w/ unk ANC lung (Infections and infestations) | 0 (0) | 1 (1)
Infection w/ unk ANC oral cavity/gums (Infections and infestations) | 1 (1) | 0 (0)
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection w/ unk ANC ungual (nails) (Infections and infestations) | 1 (1) | 1 (2)
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 3 (3) | 0 (0)
Infection-other (Infections and infestations) | 4 (5) | 3 (3)
Edema limb (General disorders) | 6 (7) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
ALT, SGPT (Metabolism and nutrition disorders) | 7 (8) | 5 (5)
AST, SGOT (Metabolism and nutrition disorders) | 5 (6) | 6 (7)
Bilirubin (Metabolism and nutrition disorders) | 4 (6) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 3 (4) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 1 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 6 (9) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nonneuropathic lower extr muscle weak (Nervous system disorders) | 1 (1) | 0 (0)
Nonneuropathic generalized weakness (Nervous system disorders) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 11 (12) | 7 (7)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 11 (11) | 5 (5)
Depression (Psychiatric disorders) | 6 (6) | 4 (5)
Neuropathy-motor (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy-sensory (Nervous system disorders) | 5 (6) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Neurologic-other (Nervous system disorders) | 9 (9) | 5 (6)
Cataract (Eye disorders) | 2 (2) | 1 (1)
Dry eye syndrome (Eye disorders) | 3 (3) | 5 (5)
Eyelid dysfunction (Eye disorders) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Double vision (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Vision-blurred (Eye disorders) | 7 (7) | 2 (2)
Vision-flashing lights/floaters (Eye disorders) | 0 (0) | 1 (1)
Ocular-other (Eye disorders) | 8 (9) | 7 (8)
Abdomen, pain (Gastrointestinal disorders) | 6 (7) | 2 (2)
Back, pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 7 (7)
Bone, pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Breast, pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Buttock, pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Chest/thoracic pain NOS (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (7)
Esophagus, pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
External ear, pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 1 (1)
Face, pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Head/headache (General disorders) | 11 (12) | 7 (7)
Joint, pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (4)
Lip, pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lymph node, pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Neck, pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Oral cavity, pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral gums, pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pain NOS (General disorders) | 2 (3) | 3 (4)
Pelvic, pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Pleura, pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin, pain (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (2)
Stomach, pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Throat/pharynx/larynx, pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vagina, pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain-other (General disorders) | 8 (8) | 8 (10)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (24) | 16 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 12 (14)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal/GU-other (Renal and urinary disorders) | 0 (0) | 1 (1)
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast volume/hypoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Irregular menses (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Sexual/Reproductive function-Other (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Flu-like syndrome (General disorders) | 3 (3) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2) | 0 (0)
Vascular-Other (Specify) (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes